CLINICAL TRIAL: NCT06748222
Title: Harnessing E-Mindfulness Approaches for Living After Breast Cancer-HEAL-ABC
Brief Title: E-Mindfulness Approaches for Living After Breast Cancer
Acronym: HEAL-ABC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NRG-CC015; R01CA282416-01 (NIH); UG1CA189867 (NIH); NCI-2024-10767 (Other: NCI)
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Depression
Keywords: Breast Cancer; Mindfulness; Meditation; Digital
MeSH Terms: conditions — Breast Neoplasms; Depression | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness (MAPs) Live Online (Experimental): Participants assigned to MAPs Live Online (MAPs LO) will be asked to attend 2-hour group sessions once a week for 6 weeks conducted live online over Zoom. Both English and Spanish language participants will be randomized to Arm 1. Sessions will be conducted on an encrypted internet connection and recorded for quality assurance and intervention fidelity. Participants who do not have a home computer, smartphone, tablet, or internet to access the Zoom sessions will have a tablet and hotspot provided by the UCLA research team. Each session provides structured lessons and guided exercises in mindfulness as well as opportunities for reflection and group discussion. Exercises include breath, body, and sound meditations; eating and walking meditations; managing pain; working with difficult thoughts and emotions; and cultivating loving kindness. Home practice is a key component of MAPs, and participants will be instructed to practice mindfulness techniques daily, beginning with 5 minutes
  Interventions: Behavioral: Mindfulness (MAPs) Live Online
- Mindfulness (MAPs) Digital App (Experimental): Participants assigned to this condition will be asked to access the MAPs App on their home computer, smartphone, or study supplied tablet over the 6-week intervention period. This will be provided by the UCLA research team. Only English language speakers will be assigned to Arm 2, as the app is currently available only in English at this time. Participants who do not have a home computer, smartphone, tablet, or internet to access the digital app will be provided with a tablet and hotspot by the UCLA research team. The MAPs App translates the content of the MAPs intervention into an app-based format, with lessons, exercises, and guided discussions from the six 2-hour sessions separated into shorter micro-sessions. The digital program is sequential with new content and exercises building on previous sessions. Lessons and other materials are gradually unlocked as participants progress through the program. Engagement with the MAPs App will be tracked to determine "dose" of the inte
  Interventions: Behavioral: Mindfulness (MAPs) Digital App
- Meditation Only Control Group (Active Comparator): The participants assigned to this condition will be provided with access to guided audio mindfulness meditations developed by the UCLA MARC (Mindfulness Awareness Research Center) and available on an app. Both English and Spanish speakers will be assigned to Arm 3, and the meditations will be available in both languages. Participants who do not have a home computer, smartphone, tablet, or internet to access the meditations will be provided with a tablet and hotspot by the UCLA research team. Use of the meditations will be tracked to determine "dose" of the intervention received.
  All three study groups will have access to the UCLA MARC mindfulness meditation app throughout the study duration out to 6 months of follow-up.
  Interventions: Behavioral: Meditation Only Control Group

INTERVENTIONS:
Behavioral: Mindfulness (MAPs) Live Online — Exercises include breath, body, and sound meditations; eating and walking meditations; managing pain; working with difficult thoughts and emotions; and cultivating loving kindness. Home practice is a key component of MAPs, and participants will be instructed to practice mindfulness techniques daily, beginning with 5 minutes daily and increasing to 20 minutes daily using guided meditations. Attendance in the group sessions and home practice will be tracked to determine "dose" of the intervention received.
  Arms: Mindfulness (MAPs) Live Online
Behavioral: Mindfulness (MAPs) Digital App — The digital program is sequential with new content and exercises building on previous sessions. Lessons and other materials are gradually unlocked as participants progress through the program. Engagement with the MAPs App will be tracked to determine "dose" of the intervention received.
  Arms: Mindfulness (MAPs) Digital App
Behavioral: Meditation Only Control Group — Use of the meditations will be tracked to determine "dose" of the intervention received.
  Arms: Meditation Only Control Group

SUMMARY:
NRG-CC015 is a prospective, randomized phase III clinical trial to evaluate the efficacy of two distinct digital approaches for delivering a mindfulness-based intervention: a live, instructor-led version delivered over Zoom (MAPs LO), and an app-based, self-paced version (MAPs App). Participants will include younger breast cancer survivors (BCS) who were diagnosed with breast cancer at or before age 50 years, have completed their primary cancer treatment (i.e., surgery, radiation, and/or chemotherapy) at least 6 months earlier, and report elevated depressive symptoms.

DETAILED DESCRIPTION:
The goal of this trial is to determine if a digital mindfulness meditation-based intervention program can improve the mental health and well-being among younger breast cancer survivors with elevated symptoms of depression. Mindfulness meditation programs provided in person have been shown to be helpful for younger breast cancer survivors. This study will compare different digital approaches for mindfulness training to see which is the most effective.

This study will also explore mediators and moderators of intervention effects, which is key for efficiently targeting psychological resources in the oncology setting and may be particularly relevant for deciding between digital intervention approaches for individual patients. Research on moderators of in-person mindfulness-based interventions (MBIs) in cancer populations suggests that patients with worse psychological functioning at study entry tend to benefit more from these interventions, with mixed effects for other predictors. It is unclear whether more distressed patients will show similar benefits in digital interventions that lack in-person check-ins and monitoring by instructors. Thus, investigators will assess baseline distress along with key demographic characteristics and social determinants of health (e.g., race, ethnicity, education, rurality) as potential moderators. With respect to mediators, emotion regulation strategies including rumination and self-kindness have been shown to mediate effects of in-person MBIs on stress and depression in cancer populations, consistent with the broader theoretical and empirical literature on mindfulness. Determining whether these factors predict and explain effects of digital MBIs, and whether these effects differ by delivery mode, is necessary for achieving optimal outcomes of these interventions. Further, investigators will collect information on the cost-effectiveness of these programs, which is critical for payors to make coverage decisions, healthcare providers and employers to make adoption decisions, and patients to make participation decisions.

ELIGIBILITY:
Inclusion Criteria:

* The participant or a legally authorized representative must provide study-specific informed consent prior to pre-entry and, for participants treated in the U.S., authorization permitting release of personal health information.
* The participant must have been greater than or equal to 18 or less than or equal to 50 years of age at the time of breast cancer diagnosis.
* The participant must have a first-time diagnosis of non-metastatic breast cancer which is Stage 0, I, II, or III.
* The participant must have a score of greater than or equal to 5 and less than or equal to 14 on the Patient Health Questionnaire-8 item (PHQ-8).
* Participants must have completed all primary breast cancer treatments at least 6 months prior to and no more than 5 years prior to registration. Note: Primary treatments include surgery, radiation therapy, adjuvant chemotherapy, targeted therapies (e.g., PARP (poly-ADP ribose polymerase) inhibitors, CDK4/6 inhibitors, TDM-1, pertuzumab, or immunotherapy). (Participants may still be taking adjuvant therapy with trastuzumab or adjuvant endocrine therapy or completing minor reconstructive surgery.)
* Participant must be able to understand, speak, read, and write in English or Spanish.
* Participant must be willing to participate in a 6-week program to receive training in mindfulness.
* Participant must be able to use a smartphone, tablet, or other digital device.
* Sex assigned at birth must be female.

Exclusion Criteria:

* Patient Health Questionnaire-8 item (PHQ-8) score of less than 5 or greater than 14 .
* Any history or current evidence of recurrent or metastatic breast cancer.
* Current or past history of another cancer. Participants with a history of only non-melanoma skin cancer or in situ cervical cancer without chemotherapy treatment would be eligible.
* Currently pregnant or planning to become pregnant in the near future.
* Participants who are enrolled in other cancer control or behavioral intervention trials that require frequent assessments or training activities.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Self-reported depressive symptoms measured-post intervention in the Mindful Awareness Practices (MAPs) live online (LO) and the meditation only (MO) groups | 2 weeks post-intervention
  The Center for Epidemiologic Studies-Depression (CES-D) score. The score is calculated as the sum of the points for all 10 items. The score range is 0-30 and a score of 10 or greater is considered depressed.
Self-reported depressive symptoms measured-post intervention in the Mindful Awareness Practices (MAPs) App and the meditation only (MO) groups | 2 weeks post-intervention
  The Center for Epidemiologic Studies-Depression (CES-D) score. The score is calculated as the sum of the points for all 10 items. The score range is 0-30 and a score of 10 or greater is considered depressed.

SECONDARY OUTCOMES:
Self-reported depressive symptoms in the Mindful Awareness Practices (MAPs) live online (LO) and the meditation only (MO) groups over time. | 3-6 months post-intervention
  The Center for Epidemiologic Studies-Depression (CES-D) score. The score is calculated as the sum of the points for all 10 items. The score range is 0-30 and a score of 10 or greater is considered depressed.
Self-reported depressive symptoms in the Mindful Awareness Practices (MAPs) App and the meditation only (MO) groups over time. | 3-6 months post-intervention
  The Center for Epidemiologic Studies-Depression (CES-D) score. The score is calculated as the sum of the points for all 10 items. The score range is 0-30 and a score of 10 or greater is considered depressed.
Self-reported fatigue symptoms in the Mindful Awareness Practices (MAPs) live online (LO) and the meditation only (MO) groups. | 6 months post-intervention
  The Patient-Reported Outcomes Measurement Information System-Short Form-Fatigue (PROMIS SF v1.0-Fatigue 7a) score. The score is calculated as the sum of the values of the response to each question (range 7-35), then rescaled into a standardized T-score with a mean of 50 and standard deviation of 10. Higher scores indicate worse fatigue than average.
Self-reported fatigue symptoms in the Mindful Awareness Practices (MAPs) App and the meditation only (MO) groups. | 6 months post-intervention
  The Patient-Reported Outcomes Measurement Information System-Short Form-Fatigue (PROMIS SF v1.0-Fatigue 7a) score. The score is calculated as the sum of the values of the response to each question (range 7-35), then rescaled into a standardized T-score with a mean of 50 and standard deviation of 10. Higher scores indicate worse fatigue than average.

CONTACTS AND LOCATIONS:
Locations (268):
- United States (266):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Marshall Cancer Center, Cameron Park, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Rush-Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Rush MD Anderson Cancer Center at Rush Lisle, Lisle, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - UI Healthcare Mission Cancer and Blood - Pella, Pella, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - UM Capital Region Medical Center, Largo, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - MyMichigan Medical Center Gratiot, Alma, Michigan
  - MyMichigan Medical Center Alpena, Alpena, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - MyMichigan Medical Center Gladwin, Gladwin, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - MyMichigan Medical Center Mount Pleasant, Mount Pleasant, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Mississippi Baptist Medical Center, Jackson, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Lake Regional Hospital, Osage Beach, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Ocean University Medical Center, Brick, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Summit Health - Florham Park Campus, Florham Park, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Mount Sinai Queens, Astoria, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Garnet Health Medical Center, Middletown, New York
  - Mount Sinai Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Cone Health MedCenter Asheboro, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Cone Health Cancer Center at Drawbridge Parkway, Greensboro, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - WellSpan Medical Oncology and Hematology, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Cancer Center Dickson City, Dickson City, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Redeemer Health, Meadowbrook, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Beaufort Memorial Hospital, Beaufort, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Inova Loudoun Hospital, Leesburg, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Richmond Community Hospital, Richmond, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Memorial Hospital of Sweetwater County, Rock Springs, Wyoming
- Puerto Rico (2):
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan